CLINICAL TRIAL: NCT00052052
Title: An Open-Label Study of the Safety and Efficacy of Subcutaneous Recombinant Interferon Gamma-1b in Patients With Idiopathic Pulmonary Fibrosis.
Brief Title: An Open-Label Study of the Safety and Efficacy of Subcutaneous Recombinant Interferon-Gamma 1b (IFN-Gamma 1b) in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InterMune (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIPF-004
Record Dates: First submitted 2003-01-21; First posted 2003-01-23 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Lung Disease; Pulmonary Fibrosis
Keywords: idiopathic pulmonary fibrosis; IPF
MeSH Terms: conditions — Lung Diseases; Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis | interventions — Interferon-gamma

INTERVENTIONS:
Drug: interferon-gamma 1b — 200 mcg, SQ, 3x per week

SUMMARY:
Study GIPF-004 is an open-label, multicenter study that will enroll approximately 250 patients who complete Protocol GIPF-001. The purpose of this study is to assess the safety and efficacy of continued IFN-gamma 1b therapy in this well-defined cohort of patients for up to 48 weeks.

ELIGIBILITY:
Male or Female

Idiopathic Pulmonary Fibrosis

20-79 years

Must have participated in the InterMune protocol GIPF-001 study.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2002-09; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
FVC, dyspnea, DLCO, A-a gradient at rest,SGRQ,survival time, use of supplemental oxygen, QOL SF-36, TLC, time to lung transplantation or death due to IPF | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Javier Szwarcberg, MD, Study Director — InterMune
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States